CLINICAL TRIAL: NCT05550714
Title: Choice of Anesthesia in Microelectrode Recording Guided Deep Brain Stimulation for Parkinson's Disease (CHAMPION)：A Randomized Controlled, Non-Inferiority Study
Brief Title: Choice of Anesthesia in Microelectrode Recording Guided Deep Brain Stimulation for Parkinson's Disease
Acronym: CHAMPION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Director of Anesthesiology Department, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xsn20220618
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: PD - Parkinson's Disease; Dexmedetomidine; Desflurane; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Anesthesia, General; Conscious Sedation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Experimental)
  Interventions: Drug: general anesthesia
- Conscious sedation (Active Comparator)
  Interventions: Drug: Conscious sedation

INTERVENTIONS:
Drug: general anesthesia — The patients did not use any preoperative sedative drugs and were given sufentanil citrate 0.1-0.2 µg/kg, cisatracurium 0.2 mg/kg and propofol 1.5-2.0 mg/kg during anesthesia induction. After the patients were unconscious, oral endotracheal intubation was performed. Anesthesiologists should continuously monitor PetCO2 and maintain PetCO2 at 30-35 mmHg. During the operation, patients are treated with remifentanil, cisatracurium, and desflurane inhalation at 0.5-1.0 minimum alveolar concentration (MAC). In the MER process, the desflurane concentration is adjusted to maintain 0.5-0.6 MAC. If the desflurane concentration needs to be adjusted to less than 0.5 MAC during MER for various reasons, remedial measures will be implemented.
  Arms: General anesthesia
Drug: Conscious sedation — A loading dose of DEX 0.5 µg/kg was infused intravenously at a constant speed within 15 min after the patients entered the operating room, and the DEX maintenance dose was infused at 0.2-0.5 µg/kg/h until the end of the first stage (deep-brain stimulation implantation) of the operation. Maintain the BIS value at 60-80.
  Other Names: asleep-awake-asleep anesthesia
  Arms: Conscious sedation

SUMMARY:
Subthalamic nucleus (STN)-deep brain stimulation (DBS) under general anesthesia has been applied to PD patients who cannot tolerate awake surgery, but general anesthesia will affect the electrical signal in microelectrode recording (MER) to some degree. This study is a prospective randomized controlled, noninferiority study, open label, endpoint outcome evaluator blinded, two-arm study. Parkinson's disease patients undergoing STN-DBS are randomly divided into a conscious sedation group (dexmedetomidine) and a general anesthesia group (desflurane). Normalized root mean square (NRMS) is used to compare the difference of neuronal activity between the two groups. The primary outcome is the percentage of high NRMS recorded by the MER signal (with the average NRMS recorded by MER after entering the STN greater than 2.0). The secondary outcomes are the NRMS, length of the STN, number of MER tracks, and differences in clinical outcomes 6 months after the operation.

DETAILED DESCRIPTION:
STN-DBS under general anesthesia has been applied to PD patients who cannot tolerate awake surgery, but general anesthesia will affect the electrical signal in microelectrode recording (MER) to some degree. At present, there are some studies on the effects of desflurane on neuronal signal amplitude and discharge characteristics during STN-DBS in PD patients but there is no definite conclusion.

This study compares the influence of MER mapping during STN-DBS and the differences in postoperative clinical outcomes between desflurane general anesthesia and conscious sedation anesthesia to explore alternative anesthesia for DBS in PD patients who cannot tolerate local anesthesia or conscious sedation and to provide feasible anesthesia techniques for the application of MER during DBS under general anesthesia.

This study is a prospective randomized controlled, noninferiority study, open label, endpoint outcome evaluator blinded, two-arm study. Parkinson's disease patients undergoing STN-DBS are randomly divided into a conscious sedation group (dexmedetomidine) and a general anesthesia group (desflurane). The primary outcome is the percentage of high NRMS recorded by the MER signal (with the average NRMS recorded by MER after entering the STN greater than 2.0), which is used to compare the differences in neuronal electrical activities between conscious sedation and general anesthesia via desflurane groups. The secondary outcomes are the NRMS, length of the subthalamic nucleus, number of MER tracks, and differences in clinical outcomes 6 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

1.50-80 years old, ASA grade II-III; 2.Bilateral STN-DBS of patients with Parkinson's disease; 3.Signed informed consent.

Exclusion Criteria:

1. Obstructive sleep apnea;
2. BMI > 30kg/m2;
3. Estimated difficult airway;
4. Severe preoperative anxiety;
5. Serious dysfunction of important organs (i.e. heart failure, renal or liver dysfunction)
6. A history of allergy to the anaesthetics.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of high-normalized root mean square (high-NRMS) recorded by the MER signal (with the average NRMS recorded by MER after entering the STN greater than 2.0). | 1 day (during MER recording)
  We will use the root mean square (RMS) value of the MER sampled signal as the main parameter for evaluating electrode position. RMS values change with the electrode properties and other external drives related to the operating room; therefore, it is crucial to normalize the RMS to comparable values. Thus, each session's RMS in a trajectory is divided by the mean RMS of the first five stable sessions in the same trajectory. This normalized RMS (NRMS) is found to be a good measure as it reflects the relative change in the total power of the signal, which elevates dramatically entering the STN.

SECONDARY OUTCOMES:
NRMS and their stratified proportions in the CS and GA groups | 1 day (during MER recording)
  We will use the root mean square (RMS) value of the MER sampled signal as the main parameter for evaluating electrode position. RMS values change with the electrode properties and other external drives related to the operating room; therefore, it is crucial to normalize the RMS to comparable values. Thus, each session's RMS in a trajectory is divided by the mean RMS of the first five stable sessions in the same trajectory. This normalized RMS (NRMS) is found to be a good measure as it reflects the relative change in the total power of the signal, which elevates dramatically entering the STN. We will stratify the mean NRMS of the two groups at the level of 0.5, and calculate the stratified proportions.
Firing rates | 1 day (during MER recording)
  The firing rates will be calculated using customized scripts developed from the Osort toolbox.
Lengths of STN(mm) | 1 day (during MER recording)
  The STN pass length is determined as the distance from entry to exit of the STN based on the significant, clear increase in baseline unit activity and FR changes unique to STN.
Total electrode path times | 1 day (during MER recording)
  Total electrode path times are the total number of paths actually selected, which can be used as an indirect indicator to judge the accuracy of positioning.
Beta band (13-30 Hz) oscillations calculated by spectrum analysis | 1 day (during MER recording)
  Power spectrum will be calculated using a discrete Fourier transform of the sampling windows to allow evaluation of change in oscillatory activity along time. Synchronized beta band (13-30 Hz) oscillations are often observed in the dorsolateral region of the STN of PD patients and are thought to play a role in the disease pathophysiology. The power of beta band will be calculated by averaging the power across the corresponding frequency band.
Proportion of intraoperative remedial measures implemented | 1 day (during MER recording)
  If the characteristic discharge activity of neurons cannot be recovered after maintaining the target anaesthetic concentration during MER, the following procedures should be implemented: ① Reduce the concentration of anaesthetics for a short time and wait for the recovery of electrical signals; ② Readjust the target position; and ③ If the STN cannot be successfully identified by MER, implant electrodes with preoperative imaging localization.
Duration of operation and MER | 1 day (during the DBS surgery)
  The operation time and MER recording time from the start to the end.
The accuracy of the DBS electrode | Within 24 hours after the operation
  The accuracy of the target location is defined by the neurosurgeon's review of the postoperative CT scan.
Clinical efficacy measured with the improvement of the United Parkinson's Disease Rating Scale (UPDRS)-III (conditions: med on/off, stim on/off) | 6 months after STN-DBS
  UPDRS -III is the standard test used by movement disorders neurologists to measure balance impairment in PD.
Clinical efficacy measured with Levodopa equivalent daily dose (LEDD) reduction | 6 months after STN-DBS
  Dopaminergic medication is converted into levodopa equivalent, which is assessed the degree of medication reduction.
Cognitive function as measured by the Mini-Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA) | At baseline and 24 hours, 2 days, 3 days and 6 months after the operation
  MMSE and MoCA will be used to assess cognitive function
Quality of life measured with the Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | 6 months after STN-DBS
  PDQ-39 will be used to assess changes in the quality of life of the patients.
The incidence of operation-related complications | Up to 6 months after randomization
  Second operation, infection, intracranial haemorrhage, etc.
The incidence of anaesthesia-related adverse events | Up to 3 days after randomization
  Nausea, vomiting and intraoperative awareness.
Surgical experience satisfaction 24 hours after the operation and DBS satisfaction 6 months after the operation evaluated by the seven-point Likert scale | 24 hours after operation for surgical experience satisfaction and 6 months after STN-DBS for DBS satisfaction
  The seven-point Likert scale will be used in the present trial. It is a questionnaire answered by the patient 24 hours after the operation. The scale reported the experience of the patient from very dissatisfied to very satisfied, as graded from 1-7.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Xie S, Shi L, Xiong W, Chen L, Li X, Tong Y, Yang W, Wang A, Zhang J, Han R. Choice of anaesthesia in microelectrode recording-guided deep-brain stimulation for Parkinson's disease (CHAMPION): study protocol for a single-centre, open-label, non-inferiority randomised controlled trial. BMJ Open. 2023 May 30;13(5):e071726. doi: 10.1136/bmjopen-2023-071726. PMID 37253497